CLINICAL TRIAL: NCT00261859
Title: Enhancing EP-Performed Alcohol Interventions in the ED
Brief Title: Enhancing Emergency Practitioner (EP)-Performed Alcohol Interventions in the Emergency Department (ED)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 0303025116; R01AA014963-01A1 (NIH)
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Harmful Drinking
Keywords: hazardous drinking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SCA (No Intervention): Standard Care with Assessment
- SCNA (No Intervention): Standard Care No Assessment
- BNI (Experimental): Brief Negotiated Interview
  Interventions: Behavioral: BNI
- EBNI (Experimental): Enhanced Brief Negotiated Interview
  Interventions: Behavioral: BNI

INTERVENTIONS:
Behavioral: BNI — behavioral- brief intervention
  Arms: BNI; EBNI

SUMMARY:
The purpose of this study is to evaluate the effectiveness of an enhanced emergency practitioner (EP) performed brief intervention (BI), namely, the Enhanced Brief Negotiation Interview (E-BNI). This includes a basic BNI performed in the ED with referral to a primary care provider, followed by a telephone booster intervention performed by trained nurses 1-month post ED visit. The E-BNI will be compared to the basic BNI (without booster), and standard care with assessments (SC-A) and without (SC-NA). In a randomized, controlled clinical trial 900 hazardous and harmful (HH) drinkers will be randomly assigned to one of the 4 conditions. We, the researchers at Yale University, will conduct cost benefit analysis of the interventions. Follow-up assessments, at 6 and 12-months, will be obtained via interactive voice response (IVR).

DETAILED DESCRIPTION:
A critical need exists to refine and test brief interventions (BI) for Emergency Department (ED) populations with hazardous and harmful (HH) drinking that can be translated into real-world settings; and to enhance the effects of these BIs so they can be maintained over time. The ED is an ideal setting for BIs, as many ED patients who exceed low-risk recommendations do not have contact with either alcohol treatment specialists or visit primary care medical practitioners. This includes a large segment of young adults ages 18-30 whose only contact with the health care system is often an ED visit. The purpose of this study is to evaluate the effectiveness of an enhanced Emergency Practitioner (EP) performed BI, namely, the Enhanced Brief Negotiation Interview (E-BNI). This includes a basic BNI performed in the ED with referral to a primary care provider, followed by a telephone booster intervention performed by trained nurses 1-month post ED visit. The E-BNI will be compared to the basic BNI (without booster), and standard care with assessments (SC-A) and without (SC-NA). In a randomized, controlled clinical trial 900 HH drinkers will be randomly assigned to one of the 4 conditions. We will conduct cost benefit analysis of the interventions. Follow-up assessments, at 6 and 12-months, will be obtained via interactive voice response (IVR).

ELIGIBILITY:
Inclusion Criteria:

* Patients, 18 years or older, who present to the adult ED at Yale-New Haven Hospital will be screened for exceeding the NIAAA criteria for low-risk drinking
* Patients may be hazardous "at-risk" drinkers who screen over the limits, but do not currently exhibit medical, social or legal problems as a result of their drinking, or they may be harmful drinkers, presenting with an alcohol associated injury or illness.

Exclusion Criteria:

Patients will be excluded for the following reasons:

* Non-English speaking;
* Alcohol dependence;
* Current enrollment in a substance abuse treatment program;
* Current ED visit for acute psychiatric complaint;
* Condition that precludes interview i.e., life threatening injury/illness;
* In police custody; or
* Inability to provide two contact numbers for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
efficacy of brief intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gail D'Onofrio, MD, MS, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital (Adult Emergency Department), New Haven, Connecticut, United States

REFERENCES:
- [Background] D'Onofrio G, Fiellin DA, Pantalon MV, Chawarski MC, Owens PH, Degutis LC, Busch SH, Bernstein SL, O'Connor PG. A brief intervention reduces hazardous and harmful drinking in emergency department patients. Ann Emerg Med. 2012 Aug;60(2):181-92. doi: 10.1016/j.annemergmed.2012.02.006. Epub 2012 Mar 28. PMID 22459448